CLINICAL TRIAL: NCT07147257
Title: A Single-Center, Randomized, Single-Blind, Single-Dose, Parallel-Group Trial to Assess the Pharmacokinetic Similarity Between CHS-1420 40 mg/0.4 mL and HUMIRA® (Adalimumab) 40 mg/0.4 mL in Healthy Chinese Adult Participants Under Fasting Conditions
Brief Title: A Trial to Assess the Pharmacokinetic Similarity Between CHS-1420 40 mg/0.4 mL and HUMIRA® (Adalimumab) 40 mg/0.4 mL in Healthy Chinese Adult Participants Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nanjing King-Friend Biochemical Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CHS-1420-10; ChiCTR2500095973 (Registry Identifier: Chinese Clinical Trial Registry)
Record Dates: First submitted 2025-08-12; First posted 2025-08-29 (Actual); Results first posted 2026-01-09 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-08

CONDITIONS: Healthy Participants
Keywords: Adalimumab; Pharmacokinetic
MeSH Terms: interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- CHS-1420 (Experimental)
  Interventions: Biological: CHS-1420
- HUMIRA® (Active Comparator)
  Interventions: Biological: HUMIRA®

INTERVENTIONS:
Biological: CHS-1420 — Dose of 40 mg will be subcutaneously administered to participants in
  Arms: CHS-1420
Biological: HUMIRA® — Dose of 40 mg will be subcutaneously administered to participants in
  Arms: HUMIRA®

SUMMARY:
A Single-Center, Randomized, Single-Blind, Single-Dose, Parallel-Group Trial to Assess the Pharmacokinetic Similarity Between CHS-1420 40 mg/0.4 mL and HUMIRA® (Adalimumab) 40 mg/0.4 mL in Healthy Chinese Adult Participants under Fasting Conditions

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide signed Informed Consent Form before the trial, and fully understand the trial content, process and possible adverse drug reactions (ADRs)
2. Able to complete the trial in compliance with the protocol
3. Participants (including males) willing to adopt effective contraceptive methods and with no pregnancy plan from 14 days before screening to 6 months after the last scheduled visit
4. Males and females between 18 and 55 years old, inclusive
5. At least 50 kg for participants, with a Body Mass Index(BMI)=Weight/ Height2 (kg/m2) between 19.0-26.0 kg/m2, inclusive
6. No history of chro nic or serious cardiac, hepatic, renal, digestive tract,nervous system, hematologic, respiratory, dermatological, mental and metabolic disorders, etc.

Exclusion Criteria:

1. With ≥ 5 cigarettes per day on average within 3 months before screening, or not able to quit smoking during the trial
2. Allergic constitution, or allergic to the drug components and its analogues; history of allergic reaction to a biological medication
3. A history of alcohol abuse (alcohol consumption of more than 14 units per week : 1 unit of alcohol = 285 mL beer, or 25 mL spirits, or 100 mL wine)
4. Blood donation or massive blood loss (> 400 mL) within 3 months before investigational products dosing; Or any blood donation plan from screening until 3 months after administration
5. History of any major surgery within the past year, or history of any surgery within the past 6 months; or any elective medical procedures, including dental procedures
6. Any history of organ transplantation
7. Medical history of tuberculosis (or suspected tuberculosis), or with a positive tuberculosis test result
8. Medical history of heart failure or other cardiac disorders which may lead to heart failure, e.g. coronary heart disease, hypertension, senile degenerative valvular disease, rheumatic valvular heart disease, dilated cardiomyopathy, acute severe myocarditis
9. Medical history of immune system disorders (e.g. systemic lupus erythematosus, multiple sclerosis, etc.), or positive results of antinuclear antibody tests
10. Medical history of recurrent or chronic infections (including transverse myelitis, optic neuritis, other demyelinating disorders, etc.), or a history of an opportunistic infection within the past year due to bacterial, mycobacterial, invasive fungal, viral, parasitic, or other opportunistic pathogens
11. History of seizure attack
12. Medication history of TNF-α blockers e.g. Adalimumab or its analogues
13. Any medication of monoclonal antibodies within the past year before investigational products dosing
14. Any usage history of prescription medicines or OTCs (especially antibiotics), or Chinese herbal medicine or health supplementary within 30 days before investigational products dosing
15. Any vaccination within 3 months before investigational products dosing, or any plan for vaccination within 3 months after investigational products administration
16. Consumption of any special diets or food items (such as grapefruit), or strenuous exercise engagement, or other factors in the opinion of investigators affecting drug absorption, distribution, metabolism and excretion within 7 days before investigational products dosing
17. Participation in other drug clinical trials within 3 months before investigational products dosing
18. Any clinically significant abnormality findings, as judged by a clinical physican, such as physical examination, vital signs, electrocardiogram and laboratory tests, as well as Chest X-ray
19. Positive results of hepatitis B surface antigen, hepatitis C antibody, and HIV antibody or syphilis
20. Consumption of chocolate or any food/beverage containing caffeine or rich in xanthine within 48 h before investigational products dosing
21. Consumption of any products containing alcohol within 48 h before investigational products dosing, or a positive result of the alcohol breath test
22. A positive result of the drug abuse test, or a history of drug abuse in the past 5 years, or intake of any narcotic drugs within 3 months prior to the trial
23. A positive result of the pregnancy test, or in lactation during screening or the test period for female participants
24. Not tolerable on venipuncture, or a history of fainting on acupuncture and/or blood
25. Special requirements and unable to follow the unified diet
26. Unable to participate in this trial for participants' own reasons
27. Other conditions in which participants are not suitable for the trial determined by investigators

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 238 (Actual)
Dates: Start 2025-02-12 (Actual); Primary Completion 2025-05-06 (Actual); Study Completion 2025-05-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Ethics Committee of Hopeshine-Minsheng Hospital of Xinzheng, Zhengzhou, China

RESULTS

PARTICIPANT FLOW:
Groups:
- CHS-1420: CHS-1420(adalimumab) at a dose of 40 mg, administered as a single subcutaneous injection, which will be performed on day 1
- HUMIRA®: Humira (adalimumab) at a dose of 40 mg, administered as a single subcutaneous injection, which will be performed on day 1
Period: Overall Study
Arm/Group | CHS-1420 | HUMIRA®
Started | 119 | 119
Completed | 118 | 116
Not Completed | 1 | 3
Not completed — Pregnancy | 1 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Drug administration failure | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | CHS-1420 | HUMIRA® | Total
Number analyzed (Participants) | 119 | 119 | 238
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 119 | 119 | 238
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: all randomized participants
  Participants
    Female | 44 | 44 | 88
    Male | 75 | 75 | 150
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: all randomized participants
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 119 | 119 | 238
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 0 | 0 | 0
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] | 23.33 (1.437) | 23.25 (1.689) | 23.29 (1.565)

OUTCOME MEASURES:

1. Primary Outcome: Areas Under the Serum Concentration Versus Time Curve Extrapolated to Infinity (AUC0-∞)
Description: pre-dose (0 h) and at 2, 4, 8, 12,24,36,48,60,72,96,120,144,168,216,288,360,528,696,864,1032,1200,1368,1536h post-dose
Time Frame: 0 to 1536 hours post-dose
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | CHS-1420 | HUMIRA®
Number analyzed (Participants) | 117 | 116
h*ng/mL | 2321566.8 (995890.41) | 2358855.5 (1038026.70)

2. Primary Outcome: The Maximum Serum Drug Concentration (Cmax)
Description: pre-dose (0 h) and at 2, 4, 8, 12,24,36,48,60,72,96,120,144,168,216,288,360,528,696,864,1032,1200,1368,1536h post-dose
Time Frame: 0 to 1536 hours post-dose
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CHS-1420 | HUMIRA®
Number analyzed (Participants) | 119 | 118
ng/mL | 3602.38 (1145.963) | 3620.75 (1489.729)

3. Secondary Outcome: Areas Under the Serum Concentration Versus Time Curve Calculated to the Last Measurable Observation (AUC0-t)
Description: pre-dose (0 h) and at 2, 4, 8, 12,24,36,48,60,72,96,120,144,168,216,288,360,528,696,864,1032,1200,1368,1536h post-dose
Time Frame: 0 to 1536 hours post-dose
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | CHS-1420 | HUMIRA®
Number analyzed (Participants) | 118 | 117
h*ng/mL | 2153350.8 (808597.63) | 2191368.0 (884277.79)

4. Secondary Outcome: Areas Under the Serum Concentration Versus Time Curve Calculated to 65 Days Postdose(AUC0-65days)
Description: pre-dose (0 h) and at 2, 4, 8, 12,24,36,48,60,72,96,120,144,168,216,288,360,528,696,864,1032,1200,1368,1536h post-dose
Time Frame: 0 to 1536 hours post-dose
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | CHS-1420 | HUMIRA®
Number analyzed (Participants) | 118 | 117
h*ng/mL | 2154968.6 (807292.73) | 2192846.0 (883361.98)

5. Secondary Outcome: The Time to Maximum Serum Concentration(Tmax)
Description: pre-dose (0 h) and at 2, 4, 8, 12,24,36,48,60,72,96,120,144,168,216,288,360,528,696,864,1032,1200,1368,1536h post-dose
Time Frame: 0 to 1536 hours post-dose
Measure: Median (Full Range); unit: h
Arm/Group | CHS-1420 | HUMIRA®
Number analyzed (Participants) | 119 | 118
h | 168.000 [36.00 to 528.00] | 156.000 [12.00 to 360.02]

6. Secondary Outcome: The Elimination Half-life (t1/2)
Description: pre-dose (0 h) and at 2, 4, 8, 12,24,36,48,60,72,96,120,144,168,216,288,360,528,696,864,1032,1200,1368,1536h post-dose
Time Frame: 0 to 1536 hours post-dose
Measure: Mean (Standard Deviation); unit: h
Arm/Group | CHS-1420 | HUMIRA®
Number analyzed (Participants) | 117 | 116
h | 240.698 (219.3439) | 238.869 (186.2289)

7. Secondary Outcome: Elimination Rate Constant (Kel)
Description: pre-dose (0 h) and at 2, 4, 8, 12,24,36,48,60,72,96,120,144,168,216,288,360,528,696,864,1032,1200,1368,1536h post-dose
Time Frame: 0 to 1536 hours post-dose
Measure: Mean (Standard Deviation); unit: 1/h
Arm/Group | CHS-1420 | HUMIRA®
Number analyzed (Participants) | 117 | 116
1/h | 0.0053 (0.0034) | 0.0050 (0.0034)

8. Secondary Outcome: Volumeof Distribution (Vd/F)
Description: pre-dose (0 h) and at 2, 4, 8, 12,24,36,48,60,72,96,120,144,168,216,288,360,528,696,864,1032,1200,1368,1536h post-dose
Time Frame: 0 to 1536 hours post-dose
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | CHS-1420 | HUMIRA®
Number analyzed (Participants) | 117 | 116
mL | 5489.1 (3152.11) | 5687.4 (3240.04)

9. Secondary Outcome: Clearance(CL/F)
Description: pre-dose (0 h) and at 2, 4, 8, 12,24,36,48,60,72,96,120,144,168,216,288,360,528,696,864,1032,1200,1368,1536h post-dose
Time Frame: 0 to 1536 hours post-dose
Measure: Mean (Standard Deviation); unit: mL/h
Arm/Group | CHS-1420 | HUMIRA®
Number analyzed (Participants) | 117 | 116
mL/h | 20.6798 (8.8808) | 20.9731 (10.7637)

10. Secondary Outcome: Immunogenicity Estimands
Description: Presence of anti-adalimumab antibodies
Time Frame: Day1 to Day 65
Measure: Count of Participants; unit: Participants
Arm/Group | CHS-1420 | HUMIRA®
Number analyzed (Participants) | 119 | 118
Participants
  ADA positive participants at 0h | 1 | 4
  baseline negative ADA participants with at least one post dose positive ADA result | 109 | 100
  No Anit-Drug Antibody Confirmed Positive Results | 9 | 14

11. Secondary Outcome: Safety Estimands
Description: Frequency of Adverse Events
Time Frame: Day1 to Day 65
Measure: Count of Participants; unit: Participants
Arm/Group | CHS-1420 | HUMIRA®
Number analyzed (Participants) | 119 | 119
Participants | 59 | 69

ADVERSE EVENTS:
Time Frame: from enrollment until end of follow-up, up to 65 days
Arm/Group | CHS-1420 | HUMIRA®
All-Cause Mortality (participants affected / at risk) | 0/119 | 0/119
Serious Adverse Events (participants affected / at risk) | 0/119 | 0/119
Other Adverse Events (participants affected / at risk) | 59/119 | 69/119
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CHS-1420 (N=119) | HUMIRA® (N=119)
Blood triglycerides increased (Investigations) | 23 | 31
Neutrophil count decreased (Investigations) | 9 | 10
Alanine aminotransferase increased (Investigations) | 9 | 8
Lymphocyte count increased (Investigations) | 3 | 7
Low density lipoprotein increased (Investigations) | 6 | 2
Aspartate aminotransferase increased (Investigations) | 4 | 4
White blood cells urine positive (Investigations) | 3 | 5
White blood cell count decreased (Investigations) | 2 | 5
Blood uric acid increased (Investigations) | 1 | 3
Total cholesterol/HDL ratio decreased (Investigations) | 2 | 1
Blood bilirubin increased (Investigations) | 0 | 3
Electrocardiogram ST-T change (Investigations) | 2 | 0
Blood creatinine increased (Investigations) | 1 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 1
Neutrophil count increased (Investigations) | 1 | 1
Platelet count increased (Investigations) | 1 | 1
Basophil count increased (Investigations) | 1 | 0
Electrocardiogram PR shortened (Investigations) | 1 | 0
Electrocardiogram Q wave abnormal (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Urinary occult blood (Investigations) | 1 | 0
Blood fibrinogen increased (Investigations) | 0 | 1
Electrocardiogram abnormal (Investigations) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 3 | 4
Anaemia (Blood and lymphatic system disorders) | 2 | 4
Proteinuria (Renal and urinary disorders) | 2 | 2
Glycosuria (Renal and urinary disorders) | 1 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Bundle branch block right (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Atrioventricular block (Cardiac disorders) | 0 | 1
Injection site erythema (General disorders) | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 2
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 2
Injury (Injury, poisoning and procedural complications) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2025-02-05): https://cdn.clinicaltrials.gov/large-docs/57/NCT07147257/Prot_000.pdf
  • Statistical Analysis Plan (2025-06-26): https://cdn.clinicaltrials.gov/large-docs/57/NCT07147257/SAP_001.pdf